CLINICAL TRIAL: NCT00852332
Title: An Open-label, Randomised, Phase II Study of Docetaxel in Combination With a Dietary Phytonutrient in First or Second Line Treatment for Patients With HER2 Negative Locally Advanced or Metastatic Breast Cancer, or Loco-regional Recurrence Not Amenable to Treatment by Surgery or Radiotherapy.
Brief Title: Docetaxel With or Without a Phytochemical in Treating Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was stopped for futility in view of the results of the anticipated analysis
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000635901; JEANP-CURRYTAX; INCA-RECF0908; EUDRACT-2008-003930-19
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer; stage IIIA breast cancer; HER2-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Curcumin; Docetaxel

ARMS (2):
- Curcumine (Experimental): With curcumin capsules
  Interventions: Dietary Supplement: Curcumin; Drug: Taxotere
- Drug taxotere only (Active Comparator): Without curcumin
  Interventions: Drug: Taxotere

INTERVENTIONS:
Dietary Supplement: Curcumin
  Arms: Curcumine
Drug: Taxotere

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Dietary supplements, such as phytochemicals, may stop or delay the development of breast cancer. It is not yet known whether giving docetaxel together with a phytochemical is more effective than giving docetaxel alone in treating patients with breast cancer.

PURPOSE: This randomized phase II trial is studying how well giving docetaxel together with a phytochemical works compared with giving docetaxel alone as first- or second-line therapy in treating patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the response rate in HER2-negative patients with locally advanced or metastatic breast cancer or locoregional breast cancer recurrence treated with docetaxel and a dietary phytochemical vs docetaxel alone.

Secondary

* To compare the overall clinical benefit rate (i.e., objective response plus stable disease) in patients treated with these regimens.
* To compare time to progression in patients treated with these regimens.
* To compare overall survival of patients treated with these regimens.
* To assess biomarkers of response in blood samples from patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to recruitment center and line of chemotherapy (first vs second line of docetaxel). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive docetaxel as in arm I. Patients also receive an oral dietary phytochemical twice on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast, meeting 1 of the following criteria:

  * Locally advanced disease
  * Documented metastatic disease without overexpression of Her2/neu

    * Must have received prior anthracycline-containing regimen as neoadjuvant, adjuvant, or first-line chemotherapy for metastatic breast cancer
  * Loco-regional recurrence not amenable to treatment by surgery or radiotherapy
* At least one measurable lesion according to RECIST criteria

  * No bone lesion only disease
* Must be a candidate for taxane-based chemotherapy
* HER2-negative disease
* No symptomatic brain metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* WHO performance status 0-2
* Life expectancy ≥ 3 months
* ANC ≥ 2,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Serum creatinine < 140 µmol/L OR creatinine clearance > 60 mL/min
* Total bilirubin ≤ upper limit of normal (ULN)
* AST and ALT ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No history of significant neurologic (i.e., peripheral neuropathy ≥ grade 2) or psychiatric disorders, including psychotic disorders, dementia, or seizures that would prohibit the understanding, observance, and giving of informed consent
* No other prior or concomitant malignancies except adequately treated carcinoma in situ of the cervix uteri, basal cell or squamous cell carcinoma of the skin, or other cancer curatively treated with surgery and/or radiotherapy
* No concurrent severe and/or uncontrolled co-morbid medical condition
* No medically unstable patients
* No uncontrolled infection
* No autoimmune disease and/or chronic active inflammation
* No psychological, familial, social, or geographical reasons that would make clinical follow-up impossible
* No malabsorption syndrome or disease significantly affecting gastrointestinal function
* No dysphagia ≥ grade 2
* No history of hypersensitivity to taxanes or known excipients, including polysorbate 80

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior major resection of the stomach or proximal small bowel
* Prior hormonal therapy as adjuvant treatment and/or treatment of metastatic disease allowed provided that the patient has progressive disease at study entry

  * Hormonal treatment must be discontinued prior to study entry
* No more than 1 prior chemotherapy regimen for metastatic disease
* More than 30 days since prior investigational drug
* More than 3 weeks since prior NSAIDs or COX_2 inhibitors
* No other concurrent anticancer therapy
* No other concurrent dietary phytonutrients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-08; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Response rate as assessed by RECIST criteria | From the date of randomization until the end of the treatment, assessed up to 21 weeks

SECONDARY OUTCOMES:
Overall clinical benefit rate as assessed by RECIST criteria | From the date of randomization until the end of the treatment, assessed up to 21 weeks
Time to progression as assessed by RECIST criteria | From date of randomization until the date of first documented progression or date of death from any cause, assessed up to 21 weeks
Overall survival as assessed by RECIST criteria | From the date of randomization until the date of death from any cause
  Evaluate overall survival (between inclusion and death whatever the cause)
Safety as assessed by NCI CTCAE v3.0 | From the date of randomization until the end of the treatment, assessed up to 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Chollet, MD, PhD, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France